CLINICAL TRIAL: NCT03183765
Title: Intralesional Measles, Mumps, Rubella (MMR) Vaccine Versus Cryotherapy in Treatment of Multiple Common and Planter Warts : a Randomized Controlled Trial
Brief Title: Intralesional Measles, Mumps, Rubella (MMR) Vaccine Versus Cryotherapy in Treatment of Multiple Common and Planter Warts
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, GAbdelsamea, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MMRVCRYO
Record Dates: First submitted 2017-06-09; First posted 2017-06-12 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Common Wart; Plantar Wart
MeSH Terms: conditions — Warts | interventions — Measles-Mumps-Rubella Vaccine; Cryotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MMR vaccine (Experimental): Measles-Mumps-Rubella Vaccine will be injected 0.5 ml into the largest wart at 2-week intervals until complete clearance was achieved or for a maximum of 3 treatments
  Interventions: Drug: Measles-Mumps-Rubella Vaccine
- Cryotherapy (Active Comparator): patients received cryotherapy with liquid nitrogen once every 2 weeks until complete clearance or for a maximum of 3 sessions
  Interventions: Procedure: cryotherapy

INTERVENTIONS:
Drug: Measles-Mumps-Rubella Vaccine — MMR vaccine will be injected 0.5 ml into the largest wart at 2-week intervals until complete clearance was achieved or for a maximum of 3 treatments.
  Response to treatment will be evaluated 1 month after the last session by decrease in the size of warts, decrease in the number of warts and photographic comparison. The clinical response was graded into complete (complete cure), partial (if there was a decrease in the size and\or a decrease in the total number of warts), and no response (no change in size and number of warts).
  Other Names: MMR
  Arms: MMR vaccine
Procedure: cryotherapy — patients received cryotherapy with liquid nitrogen once every 2 weeks until complete clearance or for a maximum of 3 sessions.Response to treatment will be evaluated 1 month after the last session by decrease in the size of warts, decrease in the number of warts and photographic comparison.
  The clinical response was graded into complete (complete cure), partial (if there was a decrease in the size and\or a decrease in the total number of warts), and no response (no change in size and number of warts).
  Arms: Cryotherapy

SUMMARY:
Warts are benign epidermal tumors caused by human papilloma virus, which are epitheliotropic non-enveloped double stranded DNA viruses. Transmission of warts occurs from direct person-to-person contact or indirectly by fomites . Warts appear in various forms including verruca vulgaris, plane, plantar, filiform, digitate and periungual.

DETAILED DESCRIPTION:
Treatment of warts is difficult for patients and physicians . Currently Available treatment options include cryosurgery, laser, electrosurgery, bleomycin, and topical keratolytic applications; many of them are painful, ineffective, costly and prone for recurrences.

Cryotherapy, which uses liquid nitrogen to freeze tissues and destroy warts, is one of the most common and effective treatments. freezing causes local irritation, leading the host to mount an immune reaction against the virus.

Immunotherapy appears to enhance virus recognition by immune system; allowing clearance of treated wart, distant warts , and helps to prevent infection .Recently, intralesional immunotherapy using different antigens such as mumps, Candida, and tuberculin has been proved effective in the treatment of warts.

The exact mechanism of action of intralesional immunotherapy is still obscure. Intralesional antigen injection probably induces strong non specific inflammatory response against the human papilloma virus-infected cells.

It has been suggested that intralesional measles mumps rubella vaccine results in regression of warts via induction of immune system.

ELIGIBILITY:
Inclusion Criteria:

* Patients should have multiple common or plantar warts.
* No concurrent systemic or topical treatment of warts

Exclusion Criteria:

* patients under 16 years old.

  • Patients with fever or signs of any inflammation or infection.
* Patients with other types of warts.
* Patients with single warts.

  * Pregnancy.
  * Lactation.
  * Immunosuppression.
  * Patients who received any other treatments for their warts in the month before starting study.
  * Past history of asthma, allergic skin disorders, meningitis or convulsions.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Cure rate | 60 days
  Assess cure rate of MMR vaccine and cryotherapy in treatment of common and planter warts (complete disappearance of lesions) one month after last session, compare efficacy of both measures.

SECONDARY OUTCOMES:
Detection of partial response to both measures | 60 days
  if there was a decrease in the size or a decrease in the total number of warts
Side effects | 60 days
  Detection of post procedure side effects such as flu like symptoms, pain , hypopigmentation.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university hospitals, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shaheen MA, Salem SA, Fouad DA, El-Fatah AA. Intralesional tuberculin (PPD) versus measles, mumps, rubella (MMR) vaccine in treatment of multiple warts: a comparative clinical and immunological study. Dermatol Ther. 2015 Jul-Aug;28(4):194-200. doi: 10.1111/dth.12230. Epub 2015 Apr 6. PMID 25847793
- [Background] Tomson N, Sterling J, Ahmed I, Hague J, Berth-Jones J. Human papillomavirus typing of warts and response to cryotherapy. J Eur Acad Dermatol Venereol. 2011 Sep;25(9):1108-11. doi: 10.1111/j.1468-3083.2010.03906.x. Epub 2010 Nov 25. PMID 21812829
- [Background] Nofal A, Nofal E, Yosef A, Nofal H. Treatment of recalcitrant warts with intralesional measles, mumps, and rubella vaccine: a promising approach. Int J Dermatol. 2015 Jun;54(6):667-71. doi: 10.1111/ijd.12480. Epub 2014 Jul 29. PMID 25070525
- [Background] Johnson SM, Roberson PK, Horn TD. Intralesional injection of mumps or Candida skin test antigens: a novel immunotherapy for warts. Arch Dermatol. 2001 Apr;137(4):451-5. PMID 11295925
- [Background] Sapp M, Bienkowska-Haba M. Viral entry mechanisms: human papillomavirus and a long journey from extracellular matrix to the nucleus. FEBS J. 2009 Dec;276(24):7206-16. doi: 10.1111/j.1742-4658.2009.07400.x. PMID 19878308
- [Background] Castellsague X, Cohet C, Puig-Tintore LM, Acebes LO, Salinas J, San Martin M, Breitscheidel L, Remy V. Epidemiology and cost of treatment of genital warts in Spain. Eur J Public Health. 2009 Jan;19(1):106-10. doi: 10.1093/eurpub/ckn127. Epub 2008 Dec 26. PMID 19112075
- [Background] Choi MH, Seo SH, Kim IH, Son SW. Comparative study on the sustained efficacy of diphencyprone immunotherapy versus cryotherapy in viral warts. Pediatr Dermatol. 2008 May-Jun;25(3):398-9. doi: 10.1111/j.1525-1470.2008.00696.x. PMID 18577059